CLINICAL TRIAL: NCT01005524
Title: A Feasibility Study for Daily Use of a Brain Computer Interface for Communication in an ICU
Brief Title: Brain Computer Interface for Communication in ICU: a Feasibility Study
Acronym: RoBIK-1
Status: Completed | Type: Observational
Sponsor: University of Versailles (Other)
Responsible Party: Principal Investigator, Djillali Annane, Head of ICU, University of Versailles
Other Study IDs: ANR-TecSan-2009; AFM2009
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Tetraplegia; Guillain-Barre Syndrome
Keywords: brain computer interface; P3Speller; P300; Event Related potential; tetraplegia; Guillain barre syndrome; Feasibility; Speed of spelling; Accuracy
MeSH Terms: conditions — Quadriplegia; Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of this study is to evaluate the usability of a system to assist verbal communication based on BCI system using the P300 wave in patients with tetraplegia who can no longer communicate because of severe engine damage (tetraplegia) and respiratory damage requiring invasive mechanical ventilation (intubation or tracheostomy) preventing verbal communication.

ELIGIBILITY:
Inclusion Criteria:

* Admitted in the ICU
* Quadriplegic and requiring mechanical ventilation (tracheostomy) 24/24h

Exclusion Criteria:

* Acute respiratory failure.
* Visual disorder
* Cognitive disorder
* Illiterate patient
* Mother tongue other than french

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Quadriplegia, also known as tetraplegia, is paralysis caused by illness or injury to a human that results in the partial or total loss of use of all of their limbs and torso; paraplegia is similar but does not affect the arms. The loss is usually sensory and motor, which means both sensation and control are lost.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de reanimation, Hopital Raymond Poincare, Garches, France

REFERENCES:
- See also: Related Info — http://www.bci2000.org
- See also: Software used for BCI — http://openvibe.inria.fr